CLINICAL TRIAL: NCT06473922
Title: Assessing Levels of Fear and Anxiety and Monitoring Wound Healing Among Patients Who Are About to Undergo Wisdom Tooth Extraction or Jaw Implant Surgery Under Local Anesthesia Versus General Anesthesia
Brief Title: Assessing Levels of Fear and Anxiety and Monitoring Wound Healing Among Patients Who Are About to Undergo Wisdom Tooth Extraction Surgery or Jaw Implant Surgery Under Local Anesthesia Versus General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Zoya Haitov Ben Zikri, Manager of the anesthesia unit, Assaf-Harofeh Medical Center
Other Study IDs: g3b8m47a
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anasthesia: Patients who are about to undergo surgery to extract wisdom teeth or no more than 3 implants in the jaw under general anesthesia in a hospital operating room.
  Interventions: Procedure: Reginal anesthesia
- Regional anesthesia: Patients who are about to undergo surgery to extract wisdom teeth or no more than 3 implants in the jaw under regional anesthesia in the dental clinic
  Interventions: Procedure: Reginal anesthesia

INTERVENTIONS:
Procedure: Reginal anesthesia — General anesthesia

SUMMARY:
Tooth extraction is one of the most common surgical procedures in dentistry. Up to 15% of the world's adult population suffers from high anxiety about dental treatments. The stress resulting from this anxiety may cause a delay in the healing and fusion of the surgical wound. Therefore, it is possible to perform this surgical tooth extraction procedure under general anesthesia.

The purpose of the present study is to assess the level of anxiety/fear and to monitor the wound healing process among patients who are about to undergo surgery to remove wisdom teeth or no more than 3 jaw implants under local anesthesia in the dental clinic compared to patients who are about to undergo the same surgery under general anesthesia.

DETAILED DESCRIPTION:
Tooth extraction is one of the most common surgical procedures in dentistry. Up to 15% of the world's adult population suffers from high anxiety about dental treatments. The stress resulting from this anxiety may cause a delay in the healing and fusion of the surgical wound. Therefore, it is possible to perform this surgical tooth extraction procedure under general anesthesia.

The purpose of the present study is to assess the level of anxiety/fear and to monitor the wound healing process among patients who are about to undergo surgery to remove wisdom teeth or no more than 3 jaw implants under local anesthesia in the dental clinic compared to patients who are about to undergo the same surgery under general anesthesia.

The various measurements of the study will include:

Level of free cortisol hormone in saliva.The levels of this hormone are correlated to the level of fear

The level of fear of pain will be measured using the Fear of Pain Questionnaire - (FPQ-III)

The level of fear of dental pain will be measured using the short version of the fear of dental pain questionnaire - FDPQ

Level of dental anxiety - will be measured using by the dental anxiety scale of The DAS Corah

. To monitor the inflammation and wound healing, the inflammatory proliferation scale (IPR) will be used to monitor the wound healing process

The study includes 5 visits:

Visit 1: 5-7 days before surgery - in the waiting room of the dental clinic. The patients will sign an informed consent form, fill out questionnaires and a saliva test will be taken from them. A clinical assessment will be conducted by the surgeon

Visit 2: on the day of surgery, in the waiting room of the dental clinic or the operating room (depending on the type of anesthesia planned). The patients will fill out questionnaires and a saliva sample will be taken from them

Visit 3: 5 days after the surgery - in the waiting room of the dental clinic The patients will fill out questionnaires and a saliva sample will be taken from them. The surgeon will report complications and complete the IPR.

Visit 4: 14 days after surgery The surgeon will complete the IPR.

Visit 5: 6 weeks after surgery The surgeon will complete the IPR.

ELIGIBILITY:
Inclusion Criteria:

Age - from ≥ 18 years, ASA 1- or 2, Signing a written informed consent before starting all procedures related to the research, Ability to cooperate with the researcher and meet the research requirements.

Exclusion Criteria:

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and females, over 18 years of age who about to undergo surgery to extract wisdom teeth or no more than 3 implants in the jaw under local anesthesia in the dental clinic or under general anesthesia in a hospital operating room.
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Level of fear | From visit 1 which will be 5-7 days before surgery to visit 5 which will be 6 weeks after surgery
  Level of fear from pain and dental fear will be monitored by questionnaireד
Wound healing | From visit 3 which will be 5 days after surgery to visit 5 which will be 6 weeks after surgery
  Will be monitored by the IPR questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bar Yehuda, PhD, Study Director — Shamir (Asaf Harofe) medical center
Locations (1):
- Shamir (Asaf Harofe) Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No